CLINICAL TRIAL: NCT05742347
Title: Efficacy of a Skin Protectant Textile for the Management of Skin Fold Conditions
Brief Title: Skin Protectant Textile Efficacy Study for Managing Skin Fold Conditions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The site sent a formal notification letter of their decision to terminate the study.
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MED-2021-DIV80-006
Record Dates: First submitted 2023-02-10; First posted 2023-02-24 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Erythema; Maceration; Lesion Skin; Skin Folds
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Intervention Model Description: A total of 46 participants were enrolled in the study -- many contributed more than one target area for a total of 82 total target areas for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DriGo SPT (Experimental): All participants will have the DriGo skin protectant textile applied to their skin fold condition.
  Interventions: Device: DriGo Skin Protectant Textile

INTERVENTIONS:
Device: DriGo Skin Protectant Textile — All participants in this study will have the DriGo skin protectant textile applied to their skin fold condition. Erythema, denudation, maceration, odor, and moisture will be assessed following application of the SPT.

SUMMARY:
This study will evaluate the efficacy of the DriGo skin protectant textile (SPT) to manage erythema, maceration, denudation, satellite lesions, pain, itching, burning, moisture, and odor associated with skin folds (henceforth together referred to as "skin fold conditions"). Participants will be patients with skin fold conditions, which will be treated with the SPT. Healthcare providers will apply the SPT to the participants' target areas. A given participant can have up to two target areas enrolled in the study. An independent licensed clinician with experience in identifying and treating skin fold conditions, will use photographs of the skin folds and other skin-on-skin contact areas (henceforth referred to as "target area[s]") to assess the status of erythema, maceration, denudation, and satellite lesions in the target areas when the SPT is first applied (Day 0), and on Days 1, 3, and 5, during SPT changes. The Principal Investigator (PI) or qualified designee will take photographs of the target areas and assess moisture and odor in these areas. Participants will provide their impressions of pain, itching and burning in the target area(s) on the same days as the skin fold condition photography. In addition, the study will include feedback from the Health Care Providers (HCPs) about the SPT and overall experience of the participants with the SPT.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age.
* Individuals who have evidence of one or more of the following skin fold conditions: erythema, maceration, denudation, satellite lesions, pain, itching, burning, moisture, and odor.
* Individuals whose treatment plan permits assessment of the skin fold condition(s) for up to six days.

Exclusion Criteria:

* Individuals whose target area(s) are being managed with topical treatments such as antibiotics, antifungals, ointments including skin protectants, anti-itch products, anoperineal dressings or absorbent pads (eg, ARD®).
* Individuals with a known allergy or sensitivity to the ingredients in the SPT, such as the fabric or H2O2, as well as the tape that may be used to secure the SPT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bryan Medical Center, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was based on the total number of target areas for review. A minimum of 80 target areas were required to complete the enrollment.
Units Other Than Participants: target areas
Period: Overall Study
Arm/Group | DriGo SPT
Started | 47; 83 target areas
Completed | 46; 82 target areas
Not Completed | 1; 1 target areas

BASELINE CHARACTERISTICS:
Population: A total of 46 participants contributing 82 target areas completed the study.
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Each participant was asked by study staff to report their age in years and this was recorded on the case report form at the time of screening.
  years | 67.61 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Each participant was asked by study staff to report which sex they identify with and this information was recorded on the case report form at the time of screening.
  Participants
    Female | 37
    Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were local to Bryan Medical Center in Lincoln Nebraska, located in the Midwest United States.
  Participants
    United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Erythema
Description: The efficacy of the SPT to improve skinfold condition of erythema over three days of treatment were assessed by third party clinicians using a 5-point Likert scales, with "0" being least severe and "4" being most severe. Data is reported as the mean and standard deviation on the scale for each timepoint.
Time Frame: day 0, day 1, day 3
Population: Individuals ≥ 18 years of age. who have evidence of one or more of the following skin fold conditions: erythema, maceration, denudation, satellite lesions, pain, itching, burning, moisture, and odor
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
units on a scale
  Day 0 | 2.15 (.82)
  Day 1 | 2.15 (0.72)
  Day 3 | .78 (.81)

2. Primary Outcome: Maceration
Description: The efficacy of the SPT to improve skinfold conditions of maceration over three days of treatment were assessed by third party clinician using a 5-point Likert scales, with "0" being least severe and "4" being most severe. Data is reported as the mean and standard deviation values from the scale for each timepoint measured.
Time Frame: day 0, day 1, day 3.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
units on a scale
  Day 0 | 0.73 (0.82)
  Day 1 | 0.49 (0.65)
  Day 3 | 0.45 (0.64)

3. Primary Outcome: Denudation
Description: The efficacy of the SPT to improve skinfold conditions denudation were assessed over 3 days by a third party clinician using a 5-point Likert scales, with "0" being least severe and "4" being most severe. Data is reported as the mean and standard deviation value on the scale for each timepoint measured.
Time Frame: day 0, day 1, and day 3.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
units on a scale
  Day 0 | 0.88 (0.84)
  Day 1 | 0.60 (0.66)
  Day 3 | 0.20 (0.44)

4. Primary Outcome: Satellite Lesions
Description: The efficacy of the SPT to improve skinfold conditions of satellite lesions were assessed by a third party clinician as absent or present each day over 5 days. Results for present lesions detected presented below. Data is reported as the percentage of participants identified with any satellite lesions.
Time Frame: 5 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
participants
  day 0 | 5
  day 1 | 5
  day 3 | 3
  day 5 | 0

5. Primary Outcome: Odor
Description: The efficacy of the SPT to improve skinfold conditions of odor over five days of treatment was assessed by a third party clinician as absent or present with values for present noted below. Data is presented as the percentage of participants identified with any odor at the target area for each timepoint measured.
Time Frame: Day 0, day 1, day 3 and day 5
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
participants
  Odor Present day 0 | 23
  Odor present day 1 | 11
  Odor present day 3 | 12
  odor present day 5 | 10

6. Secondary Outcome: Survey Responses for Moisture in the Target Area(s) on Assessment of Moisture Control.
Description: survey responses for moisture in the target area(s) on Day 0, and on Days 1, 3, and 5, during SPT changes, third party clinicians assessed the moisture as either abscent/scant or small/moderate. All other patients were coded as not able to detect. Data is presented as the percentage of participants with abscent/scant moisture at each timepoint and the percentage of participants with small/moderate moisture at each timepoint.
Time Frame: Day 0, day 1, day 3, and day 5
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
participants
  Moisture absent/scant day 0 | 15
  Moisture small/moderate day 0 | 20
  Moisture absent/scant day 1 | 13
  Moisture small/moderate day 1 | 16
  Moisture absent/scant day 3 | 15
  Moisture small/moderate day 3 | 7
  Moisture absent/scant day 5 | 10
  Moisture small/moderate day 5 | 4

7. Secondary Outcome: Assessing Patient Reported Outcomes of Discomfort (Pain, Itching, Burning) Before Dressing Change
Description: Assessing Patient reported outcomes before the dressing change - VAS score 0-100 mm with 0 being the least amount of pain and 100 being the most painful.
Time Frame: day 0, day 1, day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale - VAS score 0-100 mm
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
score on a scale - VAS score 0-100 mm
  Discomfort (Pain, Itching, or Burning) experienced before the dressing change. Day 0 | 17 (34)
  Discomfort (Pain, Itching, or Burning) experienced before the dressing change. Day 1 | 0 (23)
  Discomfort (Pain, Itching, or Burning) experienced before the dressing change. Day 3 | 0 (22)

8. Secondary Outcome: Patient Report of Pain Itching or Burning After Dressing Change Day 0, Day 1, and Day 3
Description: Assessing patient reported outcomes of discomfort (Pain, Itching, or Burning) experienced after the dressing change Patient Reported Outcomes: VAS score 0-100 mm with 0 being the least painful and 100 being the most painful
Time Frame: day 0, day 1, day3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale - VAS score 0-100 mm
Arm/Group | DriGo SPT
Number analyzed (Participants) | 46
score on a scale - VAS score 0-100 mm
  discomfort (Pain, Itching, or Burning) experienced after the dressing change Day 0 | 24.7 (32)
  discomfort (Pain, Itching, or Burning) experienced after the dressing change Day 1 | 10.6 (18)
  discomfort (Pain, Itching, or Burning) experienced after the dressing change Day 3 | 8.1 (17)

9. Secondary Outcome: Did the Product Reduce Your Discomfort Assessed at Discharge Day 5
Description: Summary Statistics of: The dressing significantly reduced discomfort (Pain, Itching, and Burning) in the skin-on-skin contact area (target area) at Day 5 with 0 being not at all and 100 being absolutely yes it helped reduce my discomfort.
Time Frame: Day 5
Population: ndividuals ≥ 18 years of age. who have evidence of one or more of the following skin fold conditions: erythema, maceration, denudation, satellite lesions, pain, itching, burning, moisture, and odor
Measure: Mean (Standard Deviation); unit: score on a scale VAS score 0-100 mm
Groups:
- Summary Statistics: Summary Statistics of: The dressing significantly reduced discomfort (Pain, Itching, and Burning) in the skin-on-skin contact area (target area) at Day 5.
Arm/Group | Summary Statistics
Number analyzed (Participants) | 46
score on a scale VAS score 0-100 mm | 98 (23)

10. Secondary Outcome: The Product Dressing Was Comfortable to Wear
Description: Summary Statistics of: The dressing was comfortable to wear at at Day 5. VAS score 0-100 mm with 0 being not at all comfortable and 100 being the most comfortable.
Time Frame: Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale - VAS score 0-100 mm
Arm/Group | Summary Statistics
Number analyzed (Participants) | 46
score on a scale - VAS score 0-100 mm | 96 (8.9)

11. Secondary Outcome: Summary Statistics of HCP - HCP Reported Ease of Use: VAS Score 0-100 mm
Description: Summary Statistics of HCP: Instructions for application of the skin protectant textile (SPT) were easy to understand. Health care practioniers (HCPs) answered a series of questions regarding the instructions for the product. Each question answered on a scale of 0-100 with 0 being negative/difficult/not likely to reccomend and 100 being positive/easy to use/likely to reccomend to others. Data is reported as the mean value for the question asked based on the scale value of 0-100. These questions were only asked of the HCP at the end of the study on day 5.
Time Frame: End of the study on day 5
Population: HCP
Measure: Mean (Standard Deviation); unit: score on a scale - VAS score 0-100 mm
Groups:
- HCP Reported Ease of Use: VAS Score 0-100 mm: Summary Statistics of HCP: Instructions for application of the skin protectant textile (SPT) were easy to understand.
  VAS score 0-100 mm
- Summary Statistics of HCP: Summary Statistics of HCP: SPT helped alleviate the skin fold conditions of my patient.
- Summary Statistics of HCP Was Easy to Apply: Summary Statistics of: SPT was easy to apply - VAS score 0-100 mm
- Summary Statistics of: I Would Recommend DriGo to Others.: Summary Statistics of: I would recommend DriGo to others. Using VAS score 0-100 mm
Arm/Group | HCP Reported Ease of Use: VAS Score 0-100 mm | Summary Statistics of HCP | Summary Statistics of HCP Was Easy to Apply | Summary Statistics of: I Would Recommend DriGo to Others.
Number analyzed (Participants) | 40 | 40 | 40 | 40
score on a scale - VAS score 0-100 mm | 93 (12) | 89 (20) | 97 (6.8) | 94 (18)

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events or severe adverse events while they were hospitalized for up to 5 days or discharge, which ever occurred first.
Groups:
- All Participants: All participants will have the DriGo skin protectant textile applied to their skin fold condition.
  DriGo Skin Protectant Textile: All participants in this study will have the DriGo skin protectant textile applied to their skin fold condition. Erythema, denudation, maceration, odor, and moisture will be assessed following application of the SPT.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT05742347/Prot_SAP_000.pdf